CLINICAL TRIAL: NCT02997930
Title: Functional Connectivity (With fMRI) as an Objective Measure of Postoperative Cognitive Function in Elderly Fracture Hip Patients
Brief Title: fMRI Connectivity in Fracture Hip Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB201601806; OCR18886 (Other: University of Florida)
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Postoperative Delirium; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications | interventions — Mental Status and Dementia Tests; DNA Replication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elderly Hip Fracture (Experimental): Postoperative assess cognitive function in elderly subjects after fracture hip surgery. Measure function connectivity and DTI (diffusion tensor imaging) via: fMRI. Subjective measures will include: Montreal Cognitive Assessment (MoCA), Digital Clock Drawing Test Command and Copy, Wide Range Achievement Test reading subtest, Hopkins Verbal Learning Test (HVLT), General Depression Scale (GDS)
  Interventions: Behavioral: fMRI; Behavioral: Montreal Cognitive Assessment (MoCA); Behavioral: Digital Clock Drawing Test Command and Copy; Behavioral: Wide Range Achievement Test reading subtest; Behavioral: Hopkins Verbal Learning Test (HVLT); Behavioral: General Depression Scale (GDS)

INTERVENTIONS:
Behavioral: fMRI — fMRI for measuring function connectivity and DTI will be done between day 2 to day 5.
Behavioral: Montreal Cognitive Assessment (MoCA) — A measure of general cognition
Behavioral: Digital Clock Drawing Test Command and Copy — A measure of current cognition using digital pen technology
Behavioral: Wide Range Achievement Test reading subtest — A measure of premorbid intellectual estimate
Behavioral: Hopkins Verbal Learning Test (HVLT) — A measure of declarative memory
Behavioral: General Depression Scale (GDS) — A measure of the of presence of depression.

SUMMARY:
The long-term goal of this study is to evaluate cognitive function preoperatively and develop techniques of intervention in the perioperative period which would optimize brain function and functional recovery following surgery.

DETAILED DESCRIPTION:
In this protocol, subjects who are anticipated to be operated for hip fracture will be studied after surgery. Brief cognitive exam will be done followed by fMRI of connectivity and diffusion tensor imaging (DTI). Connectivity (neuronal changes) and DTI (Anisotropy and mean diffusivity) data will be compared with age matched controls and correlated with subjective measures of cognition.

ELIGIBILITY:
Inclusion Criteria:

* Patients 65 years and older
* Patients who have fracture hip and are anticipated to have surgery

Exclusion Criteria:

* Patients who have contraindications for MRI like pacemaker, automatic implanted cardiac defibrillator (AICD), implanted infusion pumps etc.
* Patients who are claustrophobic
* Patients with severe cognitive impairment (who may not be able to cooperate during the cognitive exam and fMRI)

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-01-29 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
Changes between baseline and follow up visits as assessed by fMRI | Change from baseline up to 90 days
  fMRI for measuring function connectivity and DTI

SECONDARY OUTCOMES:
Changes between baseline and follow up visits as assessed by MoCA | Change from baseline up to 90 days
  A measure of general cognition
Changes between baseline and follow up visits as assessed by Digital Clock Drawing Test Command and Copy | Change from baseline up to 90 days
  a measure of current cognition using digital pen technology
Changes between baseline and follow up visits as assessed by Wide Range Achievement Test reading subtest | Change from baseline up to 90 days
  A measure of premorbid intellectual estimate
Changes between baseline and follow up visits as assessed by HVLT | Change from baseline up to 90 days
  A measure of declarative memory

CONTACTS AND LOCATIONS:
Overall Officials: Ramachandran Ramani, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No